CLINICAL TRIAL: NCT03197493
Title: Extension of Protocol 002, Carbidopa-levodopa in Neovascular Extension of Protocol 002, Carbidopa-levodopa in Neovascular AMD
Brief Title: Extension, Carbidopa-levodopa in Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Snyder, Robert W., M.D., Ph.D., P.C. (Individual)
Collaborators: Snyder Biomedical Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0003
Record Dates: First submitted 2017-06-19; First posted 2017-06-23 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Macula; Degeneration; Retina
MeSH Terms: interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: Patients who complete 3 months of escalation dose carbidopa-levodopa, will receive 9 additional months of therapy with the highest dose used in protocol 0002, carbidopa-levodopa 25-100 mg 2 tablets TID.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carbidopa/levodopa high dose (Experimental): carbidopa-levodopa 25-100 mg 2 tablets TID
  Interventions: Drug: carbidopa-levodopa 25-100 mg

INTERVENTIONS:
Drug: carbidopa-levodopa 25-100 mg — High Dose: daily oral administration 2 tablets TID Intermediate Dose: daily oral administration 1 tablet TID
  Other Names: Sinemet

SUMMARY:
This protocol is an extension of protocol 0002, Proof of Concept and Dose Ranging Study of carbidopa-levodopa in Neovascular AMD. that is a 3 month study of escalating doses of carbidopa-levodopa in neovascular AMD. This trial is a 9 month extension for patients who successfully complete protocol 0002 and wish to continue carbidopa-levodopa therapy. It will use the two higher dose regimens of protocol 0002. these will be assigned according to how well the higher dose was tolerated in protocol 0002.

DETAILED DESCRIPTION:
This extension will employ the same medications, measurements, guidelines for anti-VEGF injections and safeguards as in protocol 0002. In combination with protocol 0002, it will provide a total of 12 months of therapy with carbidopa-levodopa.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of Protocol 002.
2. A diagnosis of AMd with choroidal neovascularization (CNV) in 1 eye.
3. Normal or Dry AMD of any grade in the second eye.
4. Age 50-85 years.
5. Willingness to maintain AREDS vitamin Supplements throughout the study, or remain off of these supplements for the duration of the study, if not taking them prior to the study.
6. Informed consent at visit 1, which is also Visit 5 of study 002.

Exclusion criteria:

1. Any current use of L-DOPA containing medication or dopamine agonist medication, or any planned use of any of these agents, except for study medication, during the study;
2. Concurrent use of monoamine oxidase (MAO) inhibitors;
3. Any eye condition, disease, or history of trauma in either eye, which can impair vision, except cataract or cataract surgery;
4. BCVA worse than 20/60 in the better eye;
5. Wet AMD in the second eye;
6. Neurologic conditions which can impair vision;
7. Parkinson's Disease;
8. Significant orthostatic hypotension, defined as a drop in systolic blood pressure, immediately upon changing from the supine to standing position, of >19 mmHg, or a symptomatic drop in systolic blood pressure, immediately upon changing from the supine to standing position;
9. Significant ECG abnormalities, as judged by the Investigator;
10. Estimated glomerular filtration rate (eGFR) <20 ml/min;
11. Liver enzymes >3 X the upper limit of normal;
12. HbA1C >9.0;
13. Any other significant lab abnormalities, as judged by the Investigator.
14. Women of childbearing potential;
15. Known retinal hemorrhage;
16. Subjects who are not fluent in English.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 35 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Snyder, MD, PhD, Principal Investigator — Robert W Snyder
Locations (1):
- Robert W Snyder, MD, PhD, PC, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbidopa/Levodopa High Dose: carbidopa-levodopa 25-100 mg 2 tablets TID
  carbidopa-levodopa 25-100 mg: High Dose: daily oral administration 2 tablets TID
Period: Overall Study
Arm/Group | Carbidopa/Levodopa High Dose
Started | 35
Completed | 30
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: This population includes participants who completed NCT03022318 (naive to anti-VEGF injections at the time of enrollment) and patients who did not complete NCT03022318 but had been exposed to anti-VEGF injections before study initiation.
Arm/Group | Carbidopa/Levodopa High Dose
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 28
Age, Continuous [Mean (Full Range); unit: years] | 75 [58 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Patients naive to anti-VEGF injections at start of study [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity by ETDRS Visual Scale Testing
Description: This outcome is a measure of letters correctly identified using an Early Treatment Diabetic Retinopathy Study chart. The higher the number of letters identified, the better the participant's visual acuity.
Time Frame: From the start of the study (Visit 1) to the last completed visit, whether due to patient withdrawal, patient death or the completion of the last visit of the study (visit 12), a maximum of 9 months following a 3 month enrollment in NCT03023059.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: Change in letters (BCVA)
Groups:
- High Dose: carbidopa-levodopa 25-100 mg 2 tablets TID
  carbidopa-levodopa 25-100 mg: High Dose: daily oral administration 2 tablets TID Intermediate Dose: daily oral administration 1 tablet TID
Arm/Group | High Dose
Number analyzed (Participants) | 30
Change in letters (BCVA) | 2.7 (1.8)

2. Secondary Outcome: Number of Adverse Events Experienced
Description: Adverse events elicited by nonspecific questioning
Time Frame: Monthly for 9 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose
Number analyzed (Participants) | 30
Participants | 3

3. Secondary Outcome: Change in Central Retinal (Macular) Thickness
Description: Central retinal thickness (in microns) is measured by spectral domain-optical coherence tomography. An increase in retinal thickness is associated with disease progression. A negative value represents a decrease in retinal thickness and therefore a positive clinical outcome measure.
Time Frame: From the start of the study (Visit 1) to the last completed visit, whether due to patient withdrawal, patient death or the completion of the last visit of the study, a maximum of 9 months.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: microns
Arm/Group | High Dose
Number analyzed (Participants) | 30
microns | -18.0 (17.5)

4. Secondary Outcome: Percent Change in Retinal Fluid From Baseline
Description: Retinal fluid changes on direct retinal examination on spectral domain - optical coherence tomography. Changes in retinal fluid were compared to baseline values. A negative percentage point represents a decrease in retinal fluid and therefore a positive clinical outcome.
Time Frame: From the start of the study (Visit 1) to the last completed visit, whether due to patient withdrawal, patient death or the completion of the last visit of the study, (visit 10), a maximum of 9 months.
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: percent change
Arm/Group | High Dose
Number analyzed (Participants) | 30
percent change | -3.8 (24.8)

ADVERSE EVENTS:
Time Frame: From the start of the study (Visit 1) to the last completed visit, whether due to patient withdrawal, patient death or the completion of the last visit of the study (visit 12), a maximum of 9 months following a 3 month enrollment in NCT03023059. A total of 9 months.
Arm/Group | High Dose
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=30)
Chest pain due to torn chest muscle (Musculoskeletal and connective tissue disorders) | 1
Lightheadedness (Nervous system disorders) | 1
Malaise (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
The major limitations of our study include the small sample size and limited patient racial diversity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03197493/Prot_001.pdf